CLINICAL TRIAL: NCT01072734
Title: Role of CXCR4/CXCL12 Axis on the Control of Humoral Immunity and Auto-immunity in Lupus Patients After Influenza Vaccine Challenge
Brief Title: Auto-immunity in Lupus Patients After Influenza Vaccine
Acronym: GRIPLUP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Valerie Millul, Department Clinical Reseach of Developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P090104
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Lupus; CXCR4 on leucocytes of patients with SLE; Influenza vaccine
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Influenza, Human | interventions — Vaccines; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine group (Experimental): single group: all included patients will receive the vaccine
  Interventions: Drug: Vaccine

INTERVENTIONS:
Drug: Vaccine — Influenza vaccine
  Other Names: Influenza vaccine

SUMMARY:
Annual influenza vaccination is recommended in patients with systemic lupus erythematosus (SLE). However some concerns remain about vaccination and the risk of lupus flare

DETAILED DESCRIPTION:
SLE is a chronic autoimmune disease associated with the production of pathogenic anti-nuclear autoantibodies (ANAs) and characterized by the loss of self tolerance and the overexpression of B cells, leading to a high immunoglobulin production, 90% being autoantibodies.

There have been concerns about the safety of vaccination in patients with autoimmune diseases as it has been hypothesised that stimulation of the immune system via vaccination may lead to an increase in disease activity. Furthermore, SLE patients display a variety of immune dysfunctions which may influence their response to influenza vaccination.

Studies indicate that, although influenza vaccination in SLE may generate autoimmune phenomena, no clinically significant increase in SLE disease activity can be expected. Therefore, influenza vaccination can be considered safe in quiescent SLE, in accordance with previous reviews on this subject

The aim of this study is to evaluate if the level of CXCR4 on leucocytes of patients with SLE could be a good prognostic marker for the efficacy and the safety of influenza vaccine in SLE patients. For that purpose, we will assay in lupus patients the cellular level of CXCR4 before and after administration of influenza vaccine and correlate the expression levels of CXCR4 with: 1) the evolution of clinical and biological signs of autoimmunity and 2) the humoral immune response towards influenza. If influenza vaccine has not been associated so far with increased risk of lupus flare, it is important to determine if patients with elevated leucocytes levels of CXCR4, (due to the impact of this molecule in humoral immunity), are more at risk of vaccine side effects particularly of autoimmune origin.

ELIGIBILITY:
Inclusion criteria :

* 18 years of age and older
* informed consent signed
* LES patients who meet the American College of Rheumatology (ACR) diagnostic criteria of SLE
* Patient able to attend all visit schedule during the month following influenza vaccine administration
* Clinical examination performed prior final inclusion with results communicated to the patient

Exclusion criteria :

* For women, being pregnant or positive pregnancy test
* Positive for HCV, HIV and HBV
* Patient treated with rituximab (anti-CD20) or stopped for less than a year.
* Patient for whom a treatment majorization is suspected within the month following influenza vaccine administration.
* Hypersensitivity to active substances, eggs and to one of the vaccine components
* Other vaccinations within the last 30 days before the inclusion at J0
* Administration of blood products such as immunoglobulins within the last 90 days before J0
* Progressive cancer, cirrhoses
* Acute severe illness within the last 30 days before inclusion at J0
* Patient non affiliated to a health social security system
* Planned participation to another clinical study during the present study period
* patient deprived of freedom by an administrative or court order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The expression of CXCR4 on B cells, T cells, monocytes and granulocytes by FACS on LES patients will be measured the day of the vaccination and then 7 and 30 days post-vaccination | 7 and 30 days post-vaccination

SECONDARY OUTCOMES:
The biological signs of autoimmunity will be followed using the routine laboratory tests such as the complement exploration and the detection of total anti-nuclear antibodies detection | one year after

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CIC Vaccinologie Hopital Cochin, Paris, France

REFERENCES:
- [Derived] Launay O, Paul S, Servettaz A, Roguet G, Rozenberg F, Lucht F, Lambert C, Presles E, Goulvestre C, Meritet JF, Galtier F, Dubray C, Lebon P, Weill B, Batteux F. Control of humoral immunity and auto-immunity by the CXCR4/CXCL12 axis in lupus patients following influenza vaccine. Vaccine. 2013 Aug 2;31(35):3492-501. doi: 10.1016/j.vaccine.2013.05.095. Epub 2013 Jun 11. PMID 23764537